CLINICAL TRIAL: NCT05355051
Title: A Phase II Study of the Combination of Azacitidine and Pembrolizumab for Patients Relapsed/Refractory Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0916; NCI-2022-03778 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2022-04-25; First posted 2022-05-02 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Hodgkin's Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Azacitidine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab plus Azacitidine (Experimental): Pembrolizumab by vein over about 30 minutes every 3 weeks. Azacitidine by vein over about 60-90 minutes on Days 1-7 of each 28-day study cycle
  Interventions: Drug: Azacytidine; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Azacytidine — Given by Vein (IV)
  Other Names: 5-azacytidine; 5-aza; Vidaza™; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
Drug: Pembrolizumab — Given by Vein (IV)
  Other Names: KEYTRUDA®

SUMMARY:
This study is a Phase II single-center clinical trial designed to assess the efficacy, safety, and tolerability of pembrolizumab in combination with the 7-day regimen of azacitidine for the treatment of relapsed/refractory HL.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objectives:

• To assess the overall response rate (ORR) of Pembrolizumab in combination with azacitidine in patients with relapsed or progressed classical Hodgkin lymphoma (HL).

Secondary Objectives:

* To assess the duration of response (DOR), relapse-free survival (RFS), and overall survival (OS) of patients with refractory/relapsed HL treated with this combination.
* To assess the safety of Pembrolizumab in combination with azacitidine in children with refractory/relapsed HL.
* To assess the proportion of patients who proceed to stem cell transplantation upon achieving response with the combination of Pembrolizumab and Azacitidine regimen.

ELIGIBILITY:
Inclusion Criteria:

* HL patients with relapse or progression. Prior checkpoint inhibitors will be allowed
* Patients with relapsed HL involving extranodal sites
* HL patients who are not regarded as a candidate for high-dose, conventional chemotherapy
* Age of enrollment: Minimum age 1 year. No maximum age, study will include anyone in the pediatric/adolescent center at MD Anderson (MDA)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3 or Lansky performance status >= 50
* Adequate renal function per age unless related to the disease
* Total bilirubin < 2 x upper limit of normal (ULN) unless increase is due to Gilbert's disease
* Aspartate Aminotransferase (AST) < 3 x ULN unless considered due to lymphoma involvement
* Provision of written informed consent or assent as per MD Anderson Cancer Center (MDACC) policy for study subjects
* Females must be surgically or biologically sterile or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment and each subsequent dose
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 4 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 1 month after the last treatment
* Males need to inform the doctor right away if the partner becomes pregnant or suspects pregnancy. While in this study and for 30 days after the last treatment the patient should not donate sperm for the purposes of reproduction. He will need to use a condom while in this study and for 30 days after the last treatment

Exclusion criteria:

* Allergy to azacitidine or pembrolizumab or the drugs' components
* Active and uncontrolled comorbidities including active uncontrolled infection, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure New York Heart Association (NYHA) class III/IV, clinically significant and uncontrolled arrhythmia as judged by the treating physician
* Patients with known infection with human immunodeficiency virus (HIV) or active Hepatitis B or C
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator
* Pregnant or breastfeeding
* Has received a live vaccine within 30 days of planned start study therapy
* Current or prior use of immunosuppressive medication within 14 days prior to the first dose of pembrolizumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent
  * Steroids as premedication for hypersensitivity reactions (eg, computed tomography [CT] scan premedication)
* Active or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegener syndrome) within the past 2 years. Subjects with childhood atopy or asthma, vitiligo, alopecia, Hashimoto syndrome, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Has known active central nervous system metastases and/or carcinomatous meningitis

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the overall response rate (ORR) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David McCall, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org